CLINICAL TRIAL: NCT02375425
Title: Optimization of the ex Vivo Challenge: Reproductive Infections and Contraception
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Katherine Bunge, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO14090571
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: HIV
Keywords: BV, HSV; contraceptive; ex vivo challenge model
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- No contraceptive use: BV-/HSV- BV-/HSV+ BV+/HSV- BV+/HSV+
  Interventions: Other: no intervention
- levonorgestrel IUD: BV-/HSV- BV-/HSV+ BV+/HSV- BV+/HSV+
  Interventions: Other: no intervention
- paraguard IUD: BV-/HSV- BV-/HSV+ BV+/HSV- BV+/HSV+
  Interventions: Other: no intervention
- DMPA: BV-/HSV- BV-/HSV+ BV+/HSV- BV+/HSV+
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention-specimen collection study only

SUMMARY:
The development of surrogates to predict HIV prevention product safety and efficacy is a high priority. An ex vivo challenge model is one such promising surrogate. Colonic tissue exposed to rectally applied microbicides in vivo and then challenged with HIV in the lab showed significant reduction in HIV replication when compared to tissue exposed to placebo gel. Currently, the ex vivo challenge model for ectocervical and vaginal tissue is under development at the Dezzutti lab at the Magee Womens Research Institute in Pittsburgh, PA. Currently the Reproductive Infectious Disease Research Group is conducting a study designed to answer important questions about the ex vivo challenge model:which HIV virus is the best to use in the laboratory and what is the best indicator of HIV infection. The proposed study delineated here will investigate the effect of BV, HSV and contraceptive use on the model . There will be two arms to the study; the first will investigate the impact of HSV and BV status and the second, contraceptive use. Vaginal and cervical biopsies will be collected from participants for the ex vivo challenge model.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45
2. HIV uninfected. Note: if a woman participated in a recent research study and has an HIV test result available from that study, this will suffice provided the date of the test is within 6 months of the enrollment visit for this trial. Otherwise, the potential participant should undergo testing at the first study visit.
3. Willing and able to give informed consent to take place in the study
4. Willing to undergo a pelvic examination and genital biopsies and HIV and HSV testing
5. Willing to provide contact information
6. Agree to be sexually abstinent for two weeks beginning one week prior to the enrollment visit

Exclusion Criteria:

1. Menopausal
2. Pregnant or within 90 days of last pregnancy
3. Hysterectomy
4. Use of a diaphragm, NuvaRing or spermicide for contraception
5. Reports a course of antibiotic therapy in the 14 days prior to enrollment
6. Known history of platelet disorder or bleeding disorder
7. Participation in another microbicide or contraceptive study or a study involving cervical and/or vaginal biopsies within one month of enrollment
8. Pelvic exam findings concerning for cervicitis including abnormal cervical discharge, erythema and edema
9. Use of any spermicide or spermicide-lubricated condom within one week of enrollment.
10. Use of any internal vaginal device or product with the exception of tampons within one week of enrollment
11. Any other condition that in the opinion of the site investigator would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: non-pregnant, HIV negative, healthy 18-45 year old women
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
HIV infection of cervical and vaginal biopsies as measured by HIV-1 p24 replication by ELISA or by qPCR for HIV provirus | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bunge, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States